CLINICAL TRIAL: NCT06184230
Title: Open Label Study to Assess the ~32-Year Persistence of Hepatitis A Antibody Among Participants in the Pivotal, Double-Blind, Placebo-Controlled Efficacy Study of VAQTA (Study 023-001)
Brief Title: Persistence of Hepatitis A Antibody in Healthy Adults ~32 Years Post Vaccination.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Best Healthcare Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Study 023-Persistence
Record Dates: First submitted 2023-12-14; First posted 2023-12-28 (Actual); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: Hepatitis A
MeSH Terms: conditions — Hepatitis A | interventions — Hepatitis A Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Revaccinated at 32 Years (Other)
  Interventions: Biological: Hepatitis A Vaccine

INTERVENTIONS:
Biological: Hepatitis A Vaccine — Hepatitis A Vaccine

SUMMARY:
The goal of this clinical trial is to evaluate the persistence of Hepatitis A antibody ~32 years post vaccination in healthy adults. The questions this study will answer are: 1) how long antibody persists and 2) The immune response to an additional dose of vaccine among those with no detectable antibody. Participants will be asked to provide a blood specimen.

Those with no detectable antibody will be offered an additional dose of vaccine.

The kinetics of antibody response in this population will be summarized.

ELIGIBILITY:
Inclusion Criteria:

* Consent obtained
* Participated in original hepatitis A study in 1991
* No detectable hepatitis A antibody ~32 years after study start

Exclusion Criteria:

* Receipt of any dose of hepatitis A vaccine other than the hepatitis A vaccine used in the initial studies
* History of hepatitis A
* Receipt of blood transfusion or blood products, including immunoglobulins, within the past 6 months.
* Receipt of any vaccine within the 14 days before receipt of the additional dose of hepatitis A vaccine or scheduled to receive any vaccine within 30 days after receipt of a booster dose of vaccine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Persistence of Antibody | 32 Years
  Hepatitis A antibody

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2023-10-24): https://cdn.clinicaltrials.gov/large-docs/30/NCT06184230/Prot_ICF_000.pdf